CLINICAL TRIAL: NCT02932579
Title: Utility of Pharmacogenomic Testing and Postoperative Dental Pain Outcomes
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Study was halted permanently due to enrollment and logistic issues.
Sponsor: University of Rochester (Other)
Responsible Party: Principal Investigator, Yanfang Ren, Professor, University of Rochester
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: UofREDC; RSRB00058833 (Other: University of Rochester)
Record Dates: First submitted 2016-09-29; First posted 2016-10-13 (Estimated); Results first posted 2022-03-16 (Actual); Last update posted 2022-03-16 (Actual); Status verified 2022-03

CONDITIONS: Pain
MeSH Terms: conditions — Pain | interventions — Pharmacogenomic Testing; Ibuprofen; Acetaminophen; oxycodone-acetaminophen; Oxycodone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Standard of Care (Active Comparator): Individuals within this group will receive standard of care for postoperative dental pain secondary to extraction of impacted mandibular third molar(s)
  Interventions: Other: Pharmacogenomic Testing
- Pharmacogenomic Group (Experimental): Individuals within this group will receive pharmacogenomic testing guided prescription of pain medication for postoperative dental pain secondary to extraction of impacted mandibular third molar(s)
  Interventions: Other: Pharmacogenomic Testing; Drug: Ibuprofen; Drug: hydroxycontin/acetominophen; Drug: acetominophen; Drug: Oxycontin/acetominophen

INTERVENTIONS:
Other: Pharmacogenomic Testing — Saliva collection (5mL)
  Other Names: PGxOne Plus
Drug: Ibuprofen — 400 mg
  Arms: Pharmacogenomic Group
Drug: hydroxycontin/acetominophen — hydroxycontin 2.5 mg, acetominophen 325 mg
  Other Names: Norco
  Arms: Pharmacogenomic Group
Drug: acetominophen — 650 mg
  Arms: Pharmacogenomic Group
Drug: Oxycontin/acetominophen — 5mg Oxycontin, 325 mg acetominophen. This will be a rescue medication is the other three pain medications do not work.
  Other Names: Percoset
  Arms: Pharmacogenomic Group

SUMMARY:
Opioid analgesics are the most common postoperative pain medications used among dentists in the United States.Although these medications are highly effective in the postoperative dental pain management, not all patients optimally benefit from this therapy. Many suffer adverse consequences such as nausea, emesis, and psychomotor impairment, and there is a high prevalence of opioid prescription misuse among substance abusers within the dental patient population.

The use of non-opioid analgesics including ibuprofen and acetaminophen in the management of postoperative dental pain has demonstrated equivalent or superior analgesic effects compared to opioid analgesic therapies, typically with significantly less adverse effects.However, despite these results, dentists have encountered a high variability in the success of non-opioid analgesic responses among the postoperative dental pain population.Thus, new strategies for earlier recognition of analgesic responses for pain medications is fundamental in the field of dentistry. Therefore, this study will evaluate the clinical utility of pharmacogenomic testing in acute postoperative dental pain management among healthy adults who undergo extraction of impacted mandibular third molar.

DETAILED DESCRIPTION:
To date, the use of pharmacogenomic methods in medicine has broadened our understanding of the important role of genes and different phenotypes/genotypes that make each individual unique in pain responses, including drug biotransformation, transportation, and drug-related side effects to name a few.Thus, recognizing the genetic profile of each individual prior to the prescription of pain medication for postoperative dental pain management will be essential to provide a more effective and safer pain therapy.Additionally, we suggest that 80% of the individuals in the general population exhibit a genetic profile that influence a normal pain response to non-opioid pain therapies. Hence we postulate that the integration of a pharmacogenomic testing to guide the prescription of ibuprofen and acetaminophen, not only, could lead to improved clinical postoperative dental pain outcomes, but also, significantly reduce opioid analgesics prescriptions by dentists.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are able to read, comprehend, and sign the consent form, and willing to stay in the study unit for up to 12 hours.
* Patients who are reliable, cooperative, and of adequate intelligence to record the requested information on the questionnaire form(s).
* Women of childbearing potential who are not pregnant, as assessed by a urine pregnancy quick test on the day of the procedure, prior to surgery. Women must be using a method of birth control deemed acceptable by the investigator and continue to use this method during the duration of dosing with study medication
* Patient who develop sufficient levels of pain (rated at 50mm or more out of a 100 mm) on the DPIS within 6 hours post-surgical extraction.
* Patients who agree not to take analgesics other than protocol-defined rescue analgesics during the post-operative treatment period of 6 hours.

  * Patients who agree to refrain from alcohol and sedative consumption during the post-operative period of 6 hours.
* Patients scheduled to undergo surgical removal of 3 or more impacted third molars, at least 1 of which must be a bony mandibular impaction. In addition, the sum of the dental impaction scores must be 9 or above, carried out by investigator.

Exclusion Criteria:

Subjects with:

* Known opioids and NSAIDs allergies (or induced asthmatic attacks)
* Known history of opioid abuse
* Recent history of gastrointestinal ulceration
* History of aspirin intolerance/cross-sensitivity
* Recent myocardial disease
* Uncontrolled hypertension
* Patients receiving anticoagulation therapy
* Uncontrolled diabetes
* Pregnant women
* Immunosuppression
* Recent history of opioid or NSAID therapies
* Subjects who do not achieve a qualifying baseline pain threshold of 50mm out of 100mm on the visual analog DIPS within 6 hours of completion of surgery

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 59 (Actual)
Dates: Start 2017-07-01 (Actual); Primary Completion 2021-01-13 (Actual); Study Completion 2021-01-13 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Eastman Institute for Oral Health, Rochester, New York, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Standard of Care | Pharmacogenomic Group
Started | 33 | 26
Completed | 29 | 25
Not Completed | 4 | 1
Not completed — Withdrawal by Subject | 4 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard of Care | Pharmacogenomic Group | Total
Number analyzed (Participants) | 33 | 26 | 59
Age, Continuous [Mean (Standard Deviation); unit: years] | 23.0 (4.2) | 24.9 (4.6) | 24.0 (4.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 16 | 36
  Male | 13 | 10 | 23
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 7 | 6 | 13
  Not Hispanic or Latino | 25 | 20 | 45
  Unknown or Not Reported | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 4 | 3 | 7
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 6 | 10 | 16
  White | 18 | 12 | 30
  More than one race | 2 | 0 | 2
  Unknown or Not Reported | 3 | 1 | 4
Region of Enrollment [Number; unit: participants]
  United States | 33 | 26 | 59

OUTCOME MEASURES:

1. Primary Outcome: Mean Pain Score
Description: To compare the pain control outcomes between a single-dose of pharmacogenomics- testing-driven-prescription of ibuprofen (400mg) or acetaminophen (650mg) with those of single-dose (standard of care) of combined formulation of hydrocodone and acetaminophen (5/650mg). A visual analog scale for dental pain will be used. Scale ranges from 0-100 with 100 worse pain.
Time Frame: 6 hours
Population: subjects completed the study
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Standard of Care | Pharmacogenomic Group
Number analyzed (Participants) | 29 | 25
units on a scale | 41.9 (24.8) | 28.9 (19.4)
Statistical Analysis 1: Comparison: Standard of Care vs Pharmacogenomic Group; Test type: Superiority; p = 0.098, t-test, 2 sided; Mean Difference (Final Values) = 13.0

2. Secondary Outcome: Number of Participants That Did Not Need Opioid Analgesic Prescriptions
Description: To determine the number of patients who did not require prescribed opioid analgesic'rescue' after pharmacogenomic-guided acute postoperative dental pain management versus those taking the non-guided combined formulation of hydrocodone and acetaminophen.
Time Frame: 6 hours
Population: subjects completed the study
Measure: Count of Participants; unit: Participants
Arm/Group | Standard of Care | Pharmacogenomic Group
Number analyzed (Participants) | 29 | 25
Participants | 7 | 4
Statistical Analysis 1: Comparison: Standard of Care vs Pharmacogenomic Group; Test type: Superiority; p = 0.740, Fisher Exact; Risk Ratio (RR) = 1.38, 95% CI 2-sided [0.45 to 4.21]

ADVERSE EVENTS:
Time Frame: 6 hours after dosing
Description: any patient reported discomfort that may or may not be related to the medications during the 6 hour observation period
Arm/Group | Standard of Care | Pharmacogenomic Group
All-Cause Mortality (participants affected / at risk) | 0/29 | 0/25
Serious Adverse Events (participants affected / at risk) | 0/29 | 0/25
Other Adverse Events (participants affected / at risk) | 10/29 | 7/25
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Standard of Care (N=29) | Pharmacogenomic Group (N=25)
nausea (Gastrointestinal disorders) | 10 (10) | 7 (7)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2017-04-01): https://cdn.clinicaltrials.gov/large-docs/79/NCT02932579/Prot_SAP_000.pdf
  • Informed Consent Form (2020-06-16): https://cdn.clinicaltrials.gov/large-docs/79/NCT02932579/ICF_001.pdf